CLINICAL TRIAL: NCT04412122
Title: The Effect of Kinesio Taping and Breathing Exercises on Pain Management Applied After Benign Gynecological Abdominal Operation: A Randomized Controlled Study
Brief Title: The Effect of Kinesio Taping and Breathing Exercises on Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Sakine Yılmaz, Assistant Professor Dr, PhD, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ethic No: 2016/12/131
Record Dates: First submitted 2020-05-25; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Pain; Gas Bloat Syndrome; Defecation Disorders
Keywords: Benign gynecological changes; Postoperative pain; Kinesio taping; Breathing exercise; Nursing
MeSH Terms: conditions — Pain, Postoperative; Gas bloat syndrome | interventions — Breathing Exercises; Control Groups

STUDY DESIGN:
Intervention Model Description: After abdominal surgery, kinesio taping and breathing exercise were applied.
  Intervention Protocol of the Study Kinesio Taping (KT) Group In the study, kinesio taping method was applied immediately after the surgical operation. The tape was applied on one centimeter above and one centimeter below the incision site with a 25% tension in web cutting technique. In order to facilitate gas passing and defecation, the tape was applied around the navel in the Y shape with a 25% tension. No tension was applied to the starting and ending points of the tape. Kinesio tape remained on women for 72 hours.
  Breathing Exercises (BE) Group Before the surgery, researchers informed the women about the purpose and benefits of breathing exercises and showed the how to perform them. Breathing exercises were performed 3 times a day for 30 minutes on the first, second and third days. 15 minutes of exercises were done while sitting and in a comfortable position and 15 minutes while mobilizing.
Who Masked: Investigator
Masking Description: The data of the research were collected with personal information, postoperative follow-up and discharge risk assessment forms and Visual Analog Scale by the researcher. Pain levels of women were evaluated with Visual Analog Scale (VAS) before and after administration of the analgesic or interventions by the researcher. Data were collected on the postoperative days 0, 1, 2 and 3 during the hospital stay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kinesio Taping (Experimental): Kinesio taping is thought to remove the barriers that slow the healing process, activate neurological suppression and reduce pain (El-Refayea, El Nahasa & Ghareebb, 2016; Kamali, Sinaei & Taherkhan, 2018). Kinesio tape stimulates cutaneous mechanoreceptors. Mechanoreceptors decrease sympathetic nervous system activity and increase parasympathetic activity, which can improve intestinal control (Azam, 2017; Szczegielniak, Krajczy, Bogacz, Luniewski & Sliwinski, 2007). Kinesio taping changes skin contours and accelerates blood flow. Increased blood flow brings more oxygen and nutrients to the area. This phenomenon contributes to the natural healing process (Kafa et al., 2015).
  Interventions: Other: Kinesio Taping
- Breathing Exercise (Experimental): Breathing exercise is accepted as a key to relaxation or cooling down (El-Refayea et al., 2016). It is stated that breathing exercises reduce anxiety by preventing the transmission of pain messages to the spinal cord (Rejeh et al., 2013), reducing the catecholamine response (Rakel & Herr, 2004) and muscle tension by distracting subjects (Kelle, Güzel & Sakallı, 2016).
  Interventions: Other: Breathing Exercise
- Kinesio Taping and Breathing Exercise (Experimental): According to the application protocols, two applications were made together.
  Interventions: Other: Kinesio Taping+Breathing Exercise
- Control Group (Other): No intervention was performed to reduce pain in the control group.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Kinesio Taping — In the study, kinesio taping method was applied immediately after the surgical operation. The tape was applied on one centimeter above and one centimeter below the incision site with a 25% tension in web cutting technique (Figure 1.). In order to facilitate gas passing and defecation, the tape was applied around the navel in the Y shape with a 25% tension (Figure 2). No tension was applied to the starting and ending points of the tape. Pain level was evaluated with VAS before and after 45 minutes of tape application. Pain level was evaluated by VAS on the 1st, 2nd and 3rd postoperative day. Kinesio tape remained on women for 72 hours.
  Arms: Kinesio Taping
Other: Breathing Exercise — Before the surgery, researchers informed the women about the purpose and benefits of breathing exercises and showed the how to perform them. Breathing exercises were performed 3 times a day for 30 minutes on the first, second and third days. 15 minutes of exercises were done while sitting and in a comfortable position and 15 minutes while mobilizing. Pain levels of women were evaluated with VAS before and after 30 minutes of breathing exercises.
  Arms: Breathing Exercise
Other: Kinesio Taping+Breathing Exercise — In the study, kinesio taping method was applied immediately after the surgical operation. . Pain level was evaluated with VAS before and after 45 minutes of tape application.Breathing exercises were performed 3 times a day for 30 minutes on the first, second and third days. 15 minutes of exercises were done while sitting and in a comfortable position and 15 minutes while mobilizing. Pain levels of women were evaluated with VAS before and after 30 minutes of breathing exercises.
  Arms: Kinesio Taping and Breathing Exercise
Other: Control Group — No intervention was performed to reduce pain in the control group.
  Arms: Control Group

SUMMARY:
A randomised clinical trial in a single centre.The aim of this study is to evaluate the effect of kinesio taping and breathing exercises on pain management applied after benign gynecological abdominal operations. A total of 132 women, divided into 4 groups of 33 subjects each, were included.Women underwent gynecological abdominal operation were assigned to the groups randomly, depending on the application of two different methods of kinesio taping and breathing exercise.In randomization, a table of numbers was created, and an equal number of women were assigned to groups with four block patterns. Using kinesio taping and breathing exercise, 33 women were included in kinesio taping group (1st Group), 33 in breathing exercise group (2nd Group), and 33 in kinesio taping + breathing exercise group (3rd Group). No intervention was applied to the women in the control group (4th Group). Pain levels of women were evaluated with Visual Analog Scale (VAS) before and after administration of the interventions.

DETAILED DESCRIPTION:
Aim: The aim of this study is to evaluate the effect of kinesio taping and breathing exercises on pain management applied after benign gynecological abdominal operations.

Design-Setting: This was an experimental, randomized controlled trial. This study was conducted at the Gynecology Service of Oncology Training and Research Hospital.

Participants: A total of 132 women, divided into 4 groups of 33 subjects each, were included.

Methods: The sampling size was calculated with G*Power Ver.3.1.9.2 computer software. A total of 132 women, 33 of whom were in kinesio taping group, 33 in breathing exercise group, 33 in kinesio taping + breathing exercise group, and 33 in the control group, who matched the sampling selection criteria, were included in the study. In randomization, a table of numbers was created, and an equal number of women were assigned to groups with four block patterns. Women underwent gynecological abdominal operation were assigned to the groups randomly, depending on the application of two different methods of kinesio taping and breathing exercise. No intervention was applied to the women in the control group.

The personal information form was filled for each individual, who agreed to participate in the study, before the procedure.

Outcome Measures Pain scores of the women in all groups before, and after the procedure were evaluated by the researcher independent from each other using Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion criteria

* Women, had an abdominal operation with pfannenstiel incision due to gynecological benign changes,
* At least 18 years of age,
* Without any dermatological disease,
* Without migraines or similar chronic pain,
* Without any intestinal problem,
* Without mental disability and communication difficulties were included in the study.

Exclusion criteria

* Women, had abdominal operation due to gynecological benign changes but with a median incision,
* Had active cellulite or any other dermatological problems,
* Had deep vein thrombosis, open wounds or skin irritation, and previously had intestinal problems were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants are women.
Enrollment: 132 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 11 MONTHS
  VAS, developed by Freyd, is a scale consisting of 100-millimeter lines and used in the assessment of pain (Yaray, Akesen, Ocakolu & Aydınlı, 2011). For pain assessment using VAS, "no pain" on one end, "worst possible pain" is written on the other end of the scale and the individual shows or marks their current situation on the 100-millimeter line (Jensen, Chen, Brugger, 2003).
Postoperative follow-up form | 11 MONTHS
  Postoperative follow-up form in the study were developed by the researcher in line with the literature, and expert opinion was obtained (Gürşen, İnanoğlu, Kaya, Akbayrak & Baltacı, 2016; Hadi & Akbar Haind, 2011; Sahai Sharma, Yadav & Bindal, 2015; Stanirowski, Wunk, Cendrowski & Sawick, 2015). The postoperative follow-up form contains questions regarding the planned interventions following surgery (pain scores before and after kinesio taping and/or breathing exercises) and the postoperative recovery process (oral intake, mobilization, gas-passing, defecation time).
Discharge risk assessment form | 11 MONTHS
  Discharge risk assessment form in the study were developed by the researcher in line with the literature, and expert opinion was obtained (Gürşen, İnanoğlu, Kaya, Akbayrak & Baltacı, 2016; Hadi & Akbar Haind, 2011; Sahai Sharma, Yadav & Bindal, 2015; Stanirowski, Wunk, Cendrowski & Sawick, 2015). Discharge risk assessment form includes questions regarding the improvement of the incision site (infection, wound color, tenderness, bleeding, ecchymosis, edema) and the individual's self-perception of healing on the day of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Sakine Yılmaz, Asistant Prof, Principal Investigator — Çankırı Karatekin University; Füsun Terzioğlu, Professor, Study Director — Atılım University
Locations (1):
- Çankırı Karatekin Univesity, Çankırı, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Refayea, G.E., El Nahasa, E.M., & Ghareebb, H.O. (2016). Effect of kinesio taping therapy combined with breathing exercises on childbirth duration and labor pain: a randomized controlled trial. Bulletin of Faculty of Physical Therapy, 21(1), 23-31.
- [Background] Kamali F, Sinaei E, Taherkhani E. Comparing spinal manipulation with and without Kinesio Taping(R) in the treatment of chronic low back pain. J Bodyw Mov Ther. 2018 Apr;22(2):540-545. doi: 10.1016/j.jbmt.2017.07.008. Epub 2017 Jul 26. PMID 29861263
- [Background] Szczegielniak, J., Krajczy, M., Bogacz, K., Luniewski, J., & Sliwinski, Z. (2007). Kinesiotaping in physiotherapy after abdominal surgery. Medsportpress, 3(4), 299-307.
- [Background] Kafa N, Citaker S, Omeroglu S, Peker T, Coskun N, Diker S. Effects of kinesiologic taping on epidermal-dermal distance, pain, edema and inflammation after experimentally induced soft tissue trauma. Physiother Theory Pract. 2015;31(8):556-61. doi: 10.3109/09593985.2015.1062943. PMID 26492435
- [Background] Rejeh N, Heravi-Karimooi M, Vaismoradi M, Jasper M. Effect of systematic relaxation techniques on anxiety and pain in older patients undergoing abdominal surgery. Int J Nurs Pract. 2013 Oct;19(5):462-70. doi: 10.1111/ijn.12088. Epub 2013 May 28. PMID 24093737
- [Background] Rakel B, Herr K. Assessment and treatment of postoperative pain in older adults. J Perianesth Nurs. 2004 Jun;19(3):194-208. doi: 10.1016/j.jopan.2004.03.005. PMID 15195278
- [Background] Kelle B, Guzel R, Sakalli H. The effect of Kinesio taping application for acute non-specific low back pain: a randomized controlled clinical trial. Clin Rehabil. 2016 Oct;30(10):997-1003. doi: 10.1177/0269215515603218. Epub 2015 Aug 27. PMID 26316553
- [Background] Gursen C, Inanoglu D, Kaya S, Akbayrak T, Baltaci G. Effects of exercise and Kinesio taping on abdominal recovery in women with cesarean section: a pilot randomized controlled trial. Arch Gynecol Obstet. 2016 Mar;293(3):557-65. doi: 10.1007/s00404-015-3862-3. Epub 2015 Sep 2. PMID 26329802
- [Background] Hadi N, Hanid AA. Lavender essence for post-cesarean pain. Pak J Biol Sci. 2011 Jun 1;14(11):664-7. doi: 10.3923/pjbs.2011.664.667. PMID 22235509
- [Background] Sahai Sharma, A., Yadav, D., & Bindal, J. (2015). A study to compare healing in postoperative wounds with occlusive gauze dressing and after omitting the dressing. Journal of Medical Science and Clinical Research, 3(5), 5734-5741.
- [Background] Stanirowski PJ, Wnuk A, Cendrowski K, Sawicki W. Growth factors, silver dressings and negative pressure wound therapy in the management of hard-to-heal postoperative wounds in obstetrics and gynecology: a review. Arch Gynecol Obstet. 2015 Oct;292(4):757-75. doi: 10.1007/s00404-015-3709-y. Epub 2015 Apr 12. PMID 25864095
- [Background] Yaray O, Akesen B, Ocaklioglu G, Aydinli U. Validation of the Turkish version of the visual analog scale spine score in patients with spinal fractures. Acta Orthop Traumatol Turc. 2011;45(5):353-8. doi: 10.3944/AOTT.2011.2528. PMID 22033000
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683